CLINICAL TRIAL: NCT06168110
Title: Transcutaneous Electrical Nerve Stimulation is a Promising Novel Non-pharmacological Treatment Alternative for Mastalgia: A Randomized Clinical Trial
Brief Title: A New Treatment Option for Mastalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Volkan Genc, MD Professor, Director, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211020
Record Dates: First submitted 2023-11-10; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Mastalgia
MeSH Terms: conditions — Mastodynia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Active Comparator)
  Interventions: Device: TENS
- Sham TENS (Sham Comparator)
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Transcutaneous electrical nerve stimulation (TENS) is a non-invasive treatment method widely used for pain control

SUMMARY:
The main objective of this study is to determine the effectiveness of transcutaneous electrical nerve stimulation (TENS) treatment on pain and quality of life in mastalgia, which treatment has not yet reached a consensus.

DETAILED DESCRIPTION:
The main objective of this study is to determine the effectiveness of transcutaneous electrical nerve stimulation (TENS) treatment on pain and quality of life in mastalgia, which treatment has not yet reached a consensus. This randomized controlled clinical trial was completed with 20 women suffering from mastalgia. Patients were randomly assigned to the TENS treatment and sham application groups. Pain intensity, pain patterns and quality of life were evaluated with Breast Pain and SF-36 questionnaires before and 10 days after treatment in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mastalgia between 18 and 70 yrs old

Exclusion Criteria:

* Previous or new diagnosis of diseases that may cause extramammary mastalgia (history of previous breast surgery; inflammatory and/or tumoral breast or chest disorders such as mastitis, fibrocystic breasts, breast cancer or chest malignancies etc.)
* Having with conditions that might prevent TENS application (pacemaker, metal prosthesis, epilepsy, etc.)
* Being unable or insufficient to fill the questionnaires.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Before and 10 days after treatment
  The Breast Pain Questionnaire (BPQ), derived from the McGill Pain Questionnaire, was used to assess breast pain intensity. It is a tool that aims to evaluate the severity, pattern, location, duration and frequency of breast pain. It is calculated on the basis of Visual analog scale (VAS) and present pain intensity (PPI) scores in addition to sensory and affective component scores. Regarding the final total BPQ scores, patients' pain severity classified as mild (0-100), moderate (100-200), and severe (>200)

SECONDARY OUTCOMES:
Quality of life | Before and 10 days after treatment
  The Turkish version of the Short Form-36 version 2 (SF-36v2) was used to assess QoL before and 10 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Genç, Assoc Prof, Principal Investigator — Ankara University
Locations (1):
- Ankara Universityt School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No